CLINICAL TRIAL: NCT00648739
Title: A Phase I/II Open Label Study To Evaluate The Safety, Pharmacokinetics And Pharmacodynamics Of ALXN6000 In Patients With Relapsing Or Refractory B-Cell Chronic Lymphocytic Leukemia Or Multiple Myeloma
Brief Title: Safety and Dose Ranging Study of Samalizumab to Treat Relapsing or Refractory CLL or MM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated by the Sponsor for administrative reasons and not due to any safety concerns.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C07-003
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Multiple Myeloma
Keywords: B-cell Chronic Lymphocytic Leukemia; Leukemia; Multiple Myeloma; CD200; Anti-CD200
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Leukemia | interventions — samalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Samalizumab (Experimental): All doses of samalizumab were individualized based on the participant's body surface area in mg/m^2 based on screening height and weight. Participants were assigned to a dose cohort, ranging from 50 to 600 mg/m^2, and received a single IV dose of samalizumab. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose. If no participants enrolled into a cohort experienced a DLT, escalation to the next dose level occurred with a new cohort. If any 1 of the initial 3 participants in the cohort experienced a DLT, the cohort was expanded to at least 6 participants. Then, if less than one third of participants within the cohort experienced a DLT, escalation to the next dose level occurred with a new cohort. Dose cohorts were enrolled sequentially.
  Interventions: Drug: Samalizumab

INTERVENTIONS:
Drug: Samalizumab — Samalizumab is a humanized anti-CD200 monoclonal antibody.
  Other Names: ALXN6000

SUMMARY:
The purpose of this study was to determine the safety and maximum tolerated dose (MTD) of ALXN6000 (samalizumab) in treating relapsing or refractory B-cell chronic lymphocytic leukemia (B-CLL) or multiple myeloma (MM) and to study how samalizumab may help the immune system fight tumors that express CD200.

DETAILED DESCRIPTION:
This was an open-label multicenter study for participants with relapsing or refractory B-CLL or MM. The study was planned to be conducted in 2 parts: Part A and Part B. Both parts were to evaluate safety, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy (to the extent possible) of samalizumab in the target participant population. Part A was designed as the open-label, intravenous (IV) single dose-escalation portion of the study to determine the MTD and to assess the overall safety of different dose levels of up to 4 IV doses of samalizumab in participants with either refractory or relapsing B-CLL or MM. Initially, at least 3 participants would be enrolled into a cohort until a dose-limiting toxicity (DLT) was reached. If any 1 of the initial 3 participants in the cohort experienced a DLT, the cohort would be expanded to at least 6 participants.

After determination of the MTD in Part A, the Sponsor was to review the safety, PK, and relevant PD data to determine the dosing administration schedule for Part B. However, no participants were enrolled for Part B, as the study was terminated by the Sponsor for administrative reasons.

Participant enrollment in Cohort 7 (600 milligrams per square meter [mg/m^2] dose level), Part A, was halted after enrollment of the first participant. The study was terminated by the Sponsor for administrative reasons and not due to any safety concerns. Participants who were on study at the time of study termination were allowed to continue until the expiry date of the drug lot being used and then were followed for 30 (±1) days per protocol. The study was terminated by the Sponsor at that time. Part B of the study was not conducted.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing or Refractory B-CLL or MM
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Anticipated survival of greater than 6 months
* Female participants of childbearing potential must agree to use 2 forms of contraception
* Participants must have a standard indication for treatment of their malignancy
* Is willing and able to give written informed consent prior to any procedure not considered standard of care

Exclusion Criteria:

* Absolute neutrophil count (ANC) < 1000 x 10^9/liter (L)
* Platelet count < 50,000 x 10^9/L
* Pregnant or lactating women
* Prior history of autoimmune hemolysis requiring therapy
* Prior history of immune thrombocytopenia
* Active autoimmune disease requiring immunosuppressive therapy
* Positive Coombs' Test (neither direct or indirect)
* Ongoing corticosteroid treatment equivalent to the mineralocorticoid potency of 10 milligrams (mg) /day of prednisone, or greater, for any condition
* Prior stem cell transplantation within 4 weeks prior to enrollment
* Prior chemotherapy for the applicable malignancy within 30 days of enrollment
* Neurosurgery or cranial radiation therapy within 1 year of enrollment
* Clinically significant renal, hepatic, or cardiopulmonary disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-06-19 (Actual); Primary Completion 2010-12-14 (Actual); Study Completion 2010-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Tucson, Arizona
  - Atlanta, Georgia
  - Morristown, New Jersey
  - Durham, North Carolina

REFERENCES:
- [Derived] Mahadevan D, Lanasa MC, Farber C, Pandey M, Whelden M, Faas SJ, Ulery T, Kukreja A, Li L, Bedrosian CL, Zhang X, Heffner LT. Phase I study of samalizumab in chronic lymphocytic leukemia and multiple myeloma: blockade of the immune checkpoint CD200. J Immunother Cancer. 2019 Aug 23;7(1):227. doi: 10.1186/s40425-019-0710-1. PMID 31443741

RESULTS

PARTICIPANT FLOW:
Groups:
- Samalizumab 50 mg/m^2: Participants assigned to this dose cohort received a single intravenous (IV) dose of samalizumab 50 mg/m^2. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose.
- Samalizumab 100 mg/m^2: Participants assigned to this dose cohort received a single IV dose of samalizumab 100 mg/m^2. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose.
- Samalizumab 200 mg/m^2: Participants assigned to this dose cohort received a single IV dose of samalizumab 200 mg/m^2. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose.
- Samalizumab 300 mg/m^2: Participants assigned to this dose cohort received a single IV dose of samalizumab 300 mg/m^2. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose.
- Samalizumab 400 mg/m^2: Participants assigned to this dose cohort received a single IV dose of samalizumab 400 mg/m^2. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose.
- Samalizumab 500 mg/m^2: Participants assigned to this dose cohort received a single IV dose of samalizumab 500 mg/m^2. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose.
- Samalizumab 600 mg/m^2: Participants assigned to this dose cohort received a single IV dose of samalizumab 600 mg/m^2. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose.
Period: Overall Study
Arm/Group | Samalizumab 50 mg/m^2 | Samalizumab 100 mg/m^2 | Samalizumab 200 mg/m^2 | Samalizumab 300 mg/m^2 | Samalizumab 400 mg/m^2 | Samalizumab 500 mg/m^2 | Samalizumab 600 mg/m^2
Started | 4 | 5 | 3 | 3 | 3 | 7 | 1
Received at Least 1 Dose of Study Drug | 4 | 5 | 3 | 3 | 3 | 7 | 1
Completed | 2 | 3 | 0 | 1 | 1 | 2 | 0
Not Completed | 2 | 2 | 3 | 2 | 2 | 5 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Investigator Considered it Advisable | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Positive Human Anti-human Antibody | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Follow-up Visits Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of samalizumab.
Groups:
- Samalizumab: All doses of samalizumab were individualized based on the participant's body surface area in mg/m^2 based on screening height and weight. Participants were assigned to a dose cohort, ranging from 50 to 600 mg/m^2, and received a single IV dose of samalizumab. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose.
Arm/Group | Samalizumab
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8629 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 18
Type of Malignancy [Count of Participants; unit: Participants]
  B-Cell Chronic Lymphocytic Leukemia | 23
  Multiple Myeloma | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) Of Samalizumab
Description: The MTD was to be defined as the dose level at which less than one-third of participants experienced a dose-limiting toxicity (DLT) during the first 28 days of treatment and immediately below the dose at which at least one-third of participants experienced a DLT.
  A DLT was defined as any Grade 3 or greater toxicity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 not related to the disease under study or its sequelae that occurred in the first 28 days after dosing in Cycle 1. The NCI CTCAE grading system for the organ of involvement was used to classify severity of adverse autoimmune reactions.
Time Frame: From first dose through 10 weeks after the last dose
Population: All participants who received at least 1 dose of samalizumab.
Measure: Number; unit: mg/m^2
Arm/Group | Samalizumab
Number analyzed (Participants) | 26
mg/m^2 | NA — The MTD was not reached. The study was terminated by the Sponsor for administrative reasons and not due to any safety concerns.

2. Primary Outcome: Number Of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any event not present prior to exposure to samalizumab or any event already present that worsened in either intensity or frequency following exposure to samalizumab. A treatment-emergent serious adverse event was defined as any event that resulted in death, was immediately life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: From first dose through 10 weeks after the last dose
Population: All participants who received at least 1 dose of samalizumab.
Measure: Number; unit: participants
Groups:
- Samalizumab 50 mg/m^2: Participants assigned to this dose cohort received a single IV dose of samalizumab 50 mg/m^2. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose.
- Overall: All doses of samalizumab were individualized based on the participant's body surface area in mg/m^2 based on screening height and weight. Participants were assigned to a dose cohort, ranging from 50 to 600 mg/m^2, and received a single IV dose of samalizumab. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose.
Arm/Group | Samalizumab 50 mg/m^2 | Samalizumab 100 mg/m^2 | Samalizumab 200 mg/m^2 | Samalizumab 300 mg/m^2 | Samalizumab 400 mg/m^2 | Samalizumab 500 mg/m^2 | Samalizumab 600 mg/m^2 | Overall
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 3 | 7 | 1 | 26
participants
  At Least 1 TEAE | 4 | 5 | 3 | 3 | 3 | 6 | 1 | 25
  Treatment-emergent Serious Adverse Event | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 6
  Discontinued due to Adverse Events | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 5
  Adverse Events Leading to Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

3. Secondary Outcome: Percent Of Bound Samalizumab On B-Cell Chronic Lymphocytic Leukemia (B-CLL) Cells In Participants With B-CLL At Baseline (Predose) And Day 1 (Postdose)
Description: Bound samalizumab was detected using a monoclonal antibody (mAb) specific for samalizumab. The binding of samalizumab to CD200 on peripheral B-CLL tumor cells was evaluated in participants with B-CLL by flow cytometry and expressed as the percent of B-CLL cells bound by samalizumab. For participants with insufficient numbers of peripheral B-CLL for analysis, the samples were documented as "unevaluable" and an analysis was not performed.
Time Frame: Baseline (Predose) and Day 1 (Postdose)
Population: All participants with B-CLL who had evaluable assessments for bound samalizumab were included in the analysis. No participants with B-CLL received samalizumab at the 600 mg/m^2 dose level.
Measure: Median (Full Range); unit: percentage of B-CLL cells bound
Arm/Group | Samalizumab 50 mg/m^2 | Samalizumab 100 mg/m^2 | Samalizumab 200 mg/m^2 | Samalizumab 300 mg/m^2 | Samalizumab 400 mg/m^2 | Samalizumab 500 mg/m^2
Number analyzed (Participants) | 4 | 5 | 2 | 2 | 3 | 5
percentage of B-CLL cells bound
  Baseline (Predose) | 0.60 [0.3 to 5.9] | 0.80 [0.2 to 2.4] | 0.50 [0.3 to 0.7] | 0.60 [0.5 to 0.7] | 3.20 [1.1 to 5.7] | 1.40 [0.1 to 2.1]
  Day 1 (Postdose) | 2.50 [1.1 to 4.8] | 3.90 [0.2 to 9.5] | 28.70 [27.8 to 29.6] | 16.80 [5 to 28.6] | 13.50 [1.7 to 71.3] | 3.40 [1 to 47]

4. Secondary Outcome: Density Of B-CLL Cells Bound At Baseline (Predose) And Day 1 (Postdose)
Description: Bound samalizumab was detected using a mAb specific for samalizumab. The binding of samalizumab to CD200 on peripheral B-CLL tumor cells was evaluated in participants with B-CLL by flow cytometry and expressed as mean channel fluorescence intensity (MFI) of bound samalizumab to provide an indication of the density of bound samalizumab on target B-CLL cells. For participants with insufficient numbers of peripheral B-CLL for analysis, the samples were documented as "unevaluable" and an analysis was not performed.
Time Frame: Baseline (Predose) and Day 1 (Postdose)
Population: as for outcome 3
Measure: Median (Full Range); unit: mean channel fluorescent intensity
Arm/Group | Samalizumab 50 mg/m^2 | Samalizumab 100 mg/m^2 | Samalizumab 200 mg/m^2 | Samalizumab 300 mg/m^2 | Samalizumab 400 mg/m^2 | Samalizumab 500 mg/m^2
Number analyzed (Participants) | 4 | 5 | 2 | 2 | 3 | 5
mean channel fluorescent intensity
  Baseline (Predose) | 2.95 [1.9 to 11] | 4.10 [3.5 to 5.6] | 3.25 [3.2 to 3.3] | 2.35 [1.7 to 3] | 2.40 [1.7 to 3.4] | 1.40 [1 to 3.7]
  Day 1 (Postdose) | 3.85 [3.3 to 4.1] | 7.10 [5 to 11.1] | 17.95 [16.6 to 19.3] | 11.20 [5.6 to 16.8] | 5.80 [4.6 to 26.6] | 2.30 [1.9 to 17.6]

5. Secondary Outcome: Clinical Response Of Participants With B-CLL Following Samalizumab Dosing Using Modified NCI Working Group Response Criteria For ORR Rate
Description: Clinical responses assessed using the Modified NCI Working Group Response Criteria. Overall Response Rate (ORR)=percentage of participants who maintained best response for ≥1 month after achieving that best response and having complete response (CR), partial response (PR), nodular partial response (nPR), or stable disease (SD). CR=absence of lymphadenopathy, hepatomegaly, or splenomegaly and normal complete blood count (CBC). PR=≥50% decrease in peripheral lymphocyte count or ≥50% reduction in lymphadenopathy, hepatomegaly, or splenomegaly and normal or 50% improvement over baseline CBC. nPR=CR participants with lymphoid aggregates. Progressive disease (PD)=>50% increase for >2 lymph nodes, spleen and/or liver size, or absolute number of circulating lymphocytes; or new lymph nodes. SD=have not achieved CR, PR, or nPR or have not shown PD. Features must be exhibited for ≥1month for CR/PR. Number of participants with individual best response and ORR for each cohort is presented.
Time Frame: From first dose through 10 weeks after the last dose
Population: All participants with B-CLL who received at least 1 dose of samalizumab.
Measure: Count of Participants; unit: Participants
Groups:
- Samalizumab 300 mg/m^2: Participants assigned to this dose cohort received a single IV 300 mg/m^2 dose of samalizumab. Participants who tolerated the drug and demonstrated at least stable disease received up to 3 additional cycles of samalizumab at the same dose originally received at a minimum of 28-day intervals and beginning no sooner than 6 weeks after the initial dose.
Arm/Group | Samalizumab 50 mg/m^2 | Samalizumab 100 mg/m^2 | Samalizumab 200 mg/m^2 | Samalizumab 300 mg/m^2 | Samalizumab 400 mg/m^2 | Samalizumab 500 mg/m^2
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 3 | 5
Participants
  Progressive Disease | 1 | 1 | 0 | 0 | 1 | 2
  Partial Response | 0 | 0 | 0 | 0 | 1 | 0
  Stable Disease | 3 | 4 | 2 | 3 | 1 | 3
  Not Evaluable | 0 | 0 | 1 | 0 | 0 | 0
  ORR | 0 | 0 | 0 | 0 | 1 | 0

6. Secondary Outcome: Clinical Response Of Participants With Multiple Myeloma (MM) Following Dosing With Samalizumab
Description: Clinical responses of samalizumab were assessed using the International Myeloma Working Group Uniform Response Criteria. ORR was defined as the percentage of participants who had either stringent complete response, complete response, very good partial response, or partial response on 2 consecutive assessments made at any time before the administration of any new therapy.
  The number of participants with the individual best response and ORR for each cohort is presented.
Time Frame: From first dose through 10 weeks after the last dose
Population: All participants with MM who received at least 1 dose of samalizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Samalizumab 500 mg/m^2 | Samalizumab 600 mg/m^2
Number analyzed (Participants) | 2 | 1
Participants
  Progressive Disease | 2 | 1
  Partial Response | 0 | 0
  Stable Disease | 0 | 0
  Not Evaluable | 0 | 0
  ORR | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 (Postdose) to the end of the follow-up period (10 weeks after the last dose)
Arm/Group | Samalizumab 50 mg/m^2 | Samalizumab 100 mg/m^2 | Samalizumab 200 mg/m^2 | Samalizumab 300 mg/m^2 | Samalizumab 400 mg/m^2 | Samalizumab 500 mg/m^2 | Samalizumab 600 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/5 | 0/3 | 0/3 | 0/3 | 0/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/5 | 0/3 | 1/3 | 1/3 | 1/7 | 0/1
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 3/3 | 3/3 | 3/3 | 6/7 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Samalizumab 50 mg/m^2 (N=4) | Samalizumab 100 mg/m^2 (N=5) | Samalizumab 200 mg/m^2 (N=3) | Samalizumab 300 mg/m^2 (N=3) | Samalizumab 400 mg/m^2 (N=3) | Samalizumab 500 mg/m^2 (N=7) | Samalizumab 600 mg/m^2 (N=1)
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Samalizumab 50 mg/m^2 (N=4) | Samalizumab 100 mg/m^2 (N=5) | Samalizumab 200 mg/m^2 (N=3) | Samalizumab 300 mg/m^2 (N=3) | Samalizumab 400 mg/m^2 (N=3) | Samalizumab 500 mg/m^2 (N=7) | Samalizumab 600 mg/m^2 (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Night blindness (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 1 | 3 | 1 | 2 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral coldness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infected epidermal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood viscosity increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermabrasion (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated by the Sponsor for administrative reasons and not due to any safety concerns. Part B of the study was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes